CLINICAL TRIAL: NCT00542217
Title: Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose-Escalation Safety, Pharmacodynamics, and Pharmacokinetics Study of Intravenous Imprime PGG™ Injection in Healthy Adult Subjects
Brief Title: Phase Ia Dose-Escalation Safety, Pharmacodynamic and Pharmacokinetic Study of Imprime PGG™ Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BIOBG-CL-001
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2007-10

CONDITIONS: Healthy
Keywords: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Placebo Comparator): Single dose of 0.5 mg/kg Imprime PGG administered over 1 hr
  Interventions: Biological: Imprime PGG
- Cohort 2 (Placebo Comparator): Single dose of 1.0 mg/kg Imprime PGG administered over 1 hr
  Interventions: Biological: Imprime PGG
- Cohort 3 (Placebo Comparator): Single dose of 2.0 mg/kg Imprime PGG administered over 1 hr
  Interventions: Biological: Imprime PGG
- Cohort 4 (Placebo Comparator): Single dose of 4.0 mg/kg Imprime PGG administered over 2 hr
  Interventions: Biological: Imprime PGG
- Cohort 5 (Placebo Comparator): Single dose of 6.0 mg/kg Imprime PGG administered over 3 hr
  Interventions: Biological: Imprime PGG

INTERVENTIONS:
Biological: Imprime PGG

SUMMARY:
The purpose of this trial is to the assess the safety, pharmacodynamics, and pharmacokinetics of escalating doses of Imprime PGG™ Injection in healthy volunteers.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of a single intravenous dose of Imprime PGG versus placebo when administered to healthy adult subjects by assessing the frequency, type, and severity of treatment emergent adverse events.

The secondary objectives are:

1. to determine the pharmacodynamics of a single intravenous dose of Imprime PGG when administered to healthy adult subjects by assessing the number of subjects who experience a 15% or more increase from baseline in the percentage of neutrophils with primed CR3; and
2. to derive the pharmacokinetic profile of a single intravenous dose of Imprime PGG when administered to healthy adult subjects by assessing the plasma concentration of Imprime PGG versus time.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 to 45 years, inclusive
2. Have a body weight of 45 to 125 kg, inclusive, and a body mass index less than or equal to 30 kg/m2
3. If female, be nonpregnant and nonnursing, and if premenopausal, have a negative urine pregnancy test confirmed prior to enrollment and practicing at least two methods of birth control
4. Be healthy as determined by the investigator on the basis of medical history, the physical examination, electrocardiogram, and clinical laboratory test results
5. Have the ability to understand the requirements of the study, have provided written informed consent, and agree to abide by the study restrictions and to return for the required assessments
6. Have provided written authorization for use and disclosure of protected health information

Exclusion Criteria:

1. Have a known hypersensitivity to baker's yeast
2. Have a history of tobacco use within 3 months of the Screening Period
3. Be a known or suspected abuser of alcohol or other drugs of abuse
4. Have an active yeast infection
5. Have a positive hepatitis B, hepatitis C, or human immunodeficiency virus test during the Screening Period
6. Except as otherwise indicated, have taken any prescription medication within 14 days of study drug administration on Day 0 or over-the-counter medication, herbal preparation, or vitamins within 1 week of study drug administration on Day 0 (The following medications are exempted from this criterion: acetaminophen [maximum 3 g/day], female hormone replacement therapy, and oral contraceptives.)
7. Have participated in an investigational drug study within 30 days or five half-lives (whichever is longer) of the Screening Period
8. Have donated or lost more than a unit of blood within 30 days of the Screening Period
9. Have any clinical condition that, in the opinion of the principal investigator, warrants exclusion from the study for either a scientific, procedural, or safety perspective

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-12; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of a single intravenous dose of Imprime PGG™ Injection (Imprime PGG) versus placebo when administered to healthy adult subjects by assessing the frequency, type, and severity of adverse events. | Prospective

SECONDARY OUTCOMES:
-To determine the pharmacodynamics of a single intravenous dose of Imprime PGG by assessing the number of subjects who experience a 15% or more increase from baseline in the percentage of neutrophils with primed complement receptor 3 (CR3) | Prospective
To derive the pharmacokinetic profile of a single intravenous dose of Imprime PGG, when administered to healthy adult subjects, by assessing the plasma concentration of Imprime PGG versus time. | Prospective